CLINICAL TRIAL: NCT01391000
Title: Light Amplification by Simulated Emission Radiation Carbon Dioxide (Laser CO2) Versus Transcutaneous Electrical Stimulation (TENS) for the Reduction of Pain in Patients After Reconstruction of the Rotator Cuff. A Randomized Controlled Trial
Brief Title: Laser CO2 Versus TENS After Reconstruction of the Rotator Cuff
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0013483
Record Dates: First submitted 2011-06-15; First posted 2011-07-11 (Estimated); Results first posted 2017-08-02 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-01

CONDITIONS: Rotator Cuff Injury
Keywords: rotator cuff surgery; pain; exercise therapy
MeSH Terms: conditions — Rotator Cuff Injuries; Pain | interventions — Lasers, Gas; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laser CO2 (Experimental)
  Interventions: Procedure: LASER CO2
- TENS (Active Comparator)
  Interventions: Procedure: TENS

INTERVENTIONS:
Procedure: LASER CO2 — The therapy is performed with the patient sitting, place the unit high above the shoulder with the following indicators: through a pulsed 40 Hz, distance between device and patient 60 cm, 10x15 cm area of application, power 2W; energy between 10 and 15 J/cm2
  Arms: Laser CO2
Procedure: TENS — Transcutaneous Electrical Nerve Application of Stimulation occurs through the use of No. 3 channels (long head of biceps area (CLB), the supraspinatus muscle area, the area medial border of the scapula.
  Duration: Twenty (20) minutes, mpulsi: 70 microsec, frequency: 100 Hz, intensity: between 20 and 40 mA.
  Arms: TENS

SUMMARY:
The purpose of this study is to evaluate the most effective method between Transcutaneous Electrical Stimulation and Light Amplification by Stimulated Emission of Radiation therapy carbon dioxide therapy for pain control in the post-surgical rehabilitation of patients treated with reconstruction of the rotator cuff.

DETAILED DESCRIPTION:
To evaluate the most effective method between Transcutaneous Electrical Stimulation and Light Amplification by Stimulated Emission of Radiation therapy carbon dioxide for pain control in the post-surgical rehabilitation of patients treated with reconstruction of the rotator cuff and to evaluate, at the end of the rehabilitation period, the range of motion, the function gained and the quality of life comparatively in the two groups of patients treated with Transcutaneous Electrical Stimulation or Light Amplification by Stimulated Emission of Radiation therapy carbon dioxide therapy.

ELIGIBILITY:
Inclusion Criteria:

* subjects after surgery for rotator cuff injury of traumatic and / or degenerative

Exclusion Criteria:

* concomitant fractures of the humerus, pace-maker, diseases for which treatments are contraindicated.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-07; Primary Completion 2013-04 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberta Monesi, PT, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Bo, Italy

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Laser CO2 | TENS
Started | 35 | 35
Completed | 33 | 35
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Laser CO2 | TENS | Total
Number analyzed (Participants) | 33 | 35 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (9.2) | 61.6 (6.5) | 59.8 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 20 | 21 | 41
Number of participants with Traumatic Lesion [Count of Participants; unit: Participants] | 18 | 12 | 30

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale Mean Score
Description: To evaluate the analgesic efficacy of Light Amplification by Stimulated Emission of Radiation carbon dioxide therapy vs Transcutaneous Electrical Nerve Stimulator during the first cycle of rehabilitation through Visual Analogue Scale, calculating the mean score in values of beginning and end of daily treatment. The scale had values from 0 to 10 where zero represented no pain and 10 the worst possible pain. More than 3 means pain.
Time Frame: Change from baseline in pain at the end of the rehabilitation cycle (two weeks)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Laser CO2 | TENS
Number analyzed (Participants) | 33 | 35
units on a scale | 1.40 [0.96 to 1.84] | 1.20 [0.73 to 1.73]

2. Secondary Outcome: Constant Murley Score for Range of Motion and Shoulder Function Assessment.
Description: The Constant Murley scale had values from 0 to 100 where zero represented the worst possible range of motion and shoulder function and 100 the best.
Time Frame: Change from baseline in range of motion at the end of the rehabilitation cycle (two weeks)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Laser CO2 | TENS
Number analyzed (Participants) | 33 | 35
units on a scale | 42.12 [36.79 to 47.45] | 41.69 [36.34 to 47.04]

3. Secondary Outcome: Short Form 12-PCS for Quality of Life Assessment
Description: The SF-12 is weighted and summed to provide easily interpretable scales for physical and mental health. SF-12 score measures substantially limited physical disability, general well-being and the perception of one's state of health, (Physical Component Summary) and also measure the psychological attitude of the patient, the limitation in social and personal activities (Mental Component Summary). Physical and Mental Health Composite Scores are computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
Time Frame: Change from baseline in quality of life at the end of the rehabilitation cycle (two weeks)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Laser CO2 | TENS
Number analyzed (Participants) | 33 | 35
units on a scale | 41.07 [38.05 to 44.09] | 41.35 [38.22 to 44.47]

ADVERSE EVENTS:
Arm/Group | Laser CO2 | TENS
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/35
Other Adverse Events (participants affected / at risk) | 0/33 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No